CLINICAL TRIAL: NCT07083102
Title: Effect of Crown Material on Gingival Microbial Colonization: A Randomized Clinical Trial
Brief Title: Effect of Crown Material on Gingival Microbial Colonization
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Fatima Nasir Cheema, Effect of Crown Material on Gingival Microbial Colonization: A Randomized Clinical Trial, Pakistan Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOD/ERB/2025/77
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-06

CONDITIONS: Microbial Colonization; Missing Teeth
MeSH Terms: conditions — Communicable Diseases; Anodontia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: • Eligible participants will be randomly assigned to one of the following groups using a computer-generated sequence with allocation concealment via sealed opaque envelopes:
  * Group A: Control group
  * Group B: Full-coverage PFM crowns
  * Group C: Full-coverage Zirconia crowns
  * Single blinding: Due to the nature of the dental procedure and patient involvement in treatment planning, participants will be informed of the crown material being used (PFM or zirconia). However, they will not be informed of the specific purpose of the study (partial blinding).
  * The microbiologist conducting sample analysis will be fully blinded to participant group allocation. Additionally, the data analyst will be blinded during statistical evaluation as well.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Control group (No Intervention): Same tooth on the contra lateral side
- Group B: Full-coverage PFM crowns (Experimental): Microbial analysis will be carried out around the PFM crowns
  Interventions: Other: Experimental
- Group C: Full-coverage Zirconia crowns (Experimental): Microbial analysis will be carried out around the Full-coverage Zirconia crowns
  Interventions: Other: Experimental

INTERVENTIONS:
Other: Experimental — * Eligible participants will be randomly assigned to one of the following groups using a computer-generated sequence with allocation concealment via sealed opaque envelopes:
    * Group A: Control group
    * Group B: Full-coverage PFM crowns
    * Group C: Full-coverage Zirconia crowns
  * Baseline gingival samples will be collected with the help of sterile swab from the target tooth region prior to prosthesis placement and at the follow-up visits i.e. 1, and 3 months; both for experimental groups and control group.
  * Microbial analysis will be conducted through culture techniques to quantify CFUs and identify species.
  * Alongside, the same sample from sterile swabs will be smeared by fixating it on a microscopic slide and then Candida albicans will be stained by Periodic Acid Schiff technique, and the bacterial species using Gram staining.
  Arms: Group B: Full-coverage PFM crowns; Group C: Full-coverage Zirconia crowns

SUMMARY:
* Prior approval from SOD ethical committee has been received.
* All patients presenting to the General OPD of School of Dentistry, Islamabad will be screened. Those patients who fulfill the criteria will be referred to the Prosthodontics department.
* The patients will undergo detailed history and oral examination after informed consent (Annexure-A). Patients will undergo radiographic investigation and based on this information they will be selected for the study according to the exclusion and inclusion criteria.
* Eligible participants will be randomly assigned to one of the following groups using a computer-generated sequence with allocation concealment via sealed opaque envelopes:

  * Group A: Control group
  * Group B: Full-coverage PFM crowns
  * Group C: Full-coverage Zirconia crowns
* Baseline gingival samples will be collected with the help of sterile swab from the target tooth region prior to prosthesis placement and at the follow-up visits i.e. 1, and 3 months; both for experimental groups and control group.
* Microbial analysis will be conducted through culture techniques to quantify CFUs and identify species.
* A summary of the micro-organisms, their incubation media, temperature and time is presented in the following table:

Table 1: Summary of the micro-organisms, their incubation media, temperature and time Micro-organism Growth Media Temperature Incubation time Candida albicans Saboraud Agar 370C 24-48 hours Streptococcus mutans BHI broth 370C 24-48 hours Staphylococcus aureus BHI broth 370C 24-48 hours Porphyromonas gingivalis BHI broth 370C 18-24 hours

* Alongside, the same sample from sterile swabs will be smeared by fixating it on a microscopic slide and then Candida albicans will be stained by Periodic Acid Schiff technique, and the bacterial species using Gram staining.
* All participants will receive standardized verbal and written instructions oral hygiene instructions to control for hygiene-related variation

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 to 50 years.
* Both male and female patients will be selected.
* Good oral hygiene (Defined as a plaque index score ≤ 1 across all assessed surfaces and no visible calculus deposits)
* Dentate patients require fixed prostheses for the first time on mandibular pre-molars and molars.
* Patient with no history of any dental and bony pathosis (cysts, cancerous lesion).

Exclusion Criteria:

* Untreated periodontal diseases
* Xerostomia
* Pregnancy, lactation
* Smokers
* Individuals with systemic conditions like diabetes and immunosuppressive diseases

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Quantitative change in gingival microbial count (CFU/ml) for each microorganism over time. | 3 months

SECONDARY OUTCOMES:
Comparative analysis of microbial colonization trends between PFM and Zirconia crown groups | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dentistry, SZAMBU, Islamabad, Federal, Pakistan